CLINICAL TRIAL: NCT04344067
Title: The Effect of Far Infrared Therapy on Peritoneal Function of CAPD Patients
Brief Title: Far Infrared Therapy on Peritoneal Function of CAPD Patients
Acronym: CAPD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-09-002B
Record Dates: First submitted 2020-03-19; First posted 2020-04-14 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: End-stage Renal Disease
Keywords: Peritoneal Dialysis; Far Infrared Therapy
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: Participants are assigned to either the control group or the treatment (far infrared therapy) group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention)
- Far Infrared Therapy Group (Experimental): In this study, the top radiator of the far infrared emitter was set at a height of 25 cm above the umbilicus with a treatment time of 40 minutes during the initial 1 hour of both the first daily and the last night-time indwelling dialysate of each daily regular peritoneal dialysis regimen.
  Interventions: Device: Far Infrared Therapy

INTERVENTIONS:
Device: Far Infrared Therapy — The WSTM TY101 FIR emitter (WS Far Infrared Medical Technology Co., Ltd., Taipei, Taiwan) was used to conduct FIR therapy in this study. The electrified ceramic plates of the emitter generated electromagnetic waves with wavelengths in the range between 3 and 25 μm (a peak between 5 to 6 μm). The irradiating power density is 10 and 20 milliwatt (mw) /cm2 when the top radiator was set at a distance of 30 and 20 cm above the skin surface respectively.
  Arms: Far Infrared Therapy Group

SUMMARY:
For patients with end-stage renal disease, peritoneal dialysis (PD) has been proven to be an alternative choice compared to hemodialysis as a type of maintenance renal replacement therapy. Despite this, long-term PD is associated with structural membrane changes that are believed to contribute to alterations in solute transport and loss of ultrafiltration. Previous studies have proven that far-infrared (FIR) therapy may improve not only the arteriovenous fistula patency in hemodialysis patients but also abdominal discomfort due to encapsulating peritoneal sclerosis in PD patients. Since there is little information concerning this issue, this study was conducted in order to evaluate the possible effects of FIR therapy on the peritoneal function of patients receiving continuous ambulatory peritoneal dialysis (CAPD). The objective of this study is to evaluate the effect of FIR therapy on the peritoneal function, protein loss, and ultrafiltration capacity of CAPD patients.

DETAILED DESCRIPTION:
A total of 100 CAPD patients will be enrolled in this study, including 50 in treatment group who will receive FIR therapy for 6 months and 50 in control group. Many parameters of blood and urine samples as well as ultrafiltration amount, dialysate urea nitrogen, creatinine, Na+, K+, total protein, CA-125, and glucose degradation product (GDP) for the dialysate effluent of not only the first and last exchanges but also the total exchanges of daily PD regimen will be measured for both groups at day 1 and 6th month. However, only the FIR group will receive tests of blood, urine and dialysate on day 2. The significance of the study is that patients might benefit from the prophylactic therapeutic effects of FIR therapy, leading to the reduction of the hospitalization costs and the need for interventional procedures in CAPD patient care in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* Chronic peritoneal dialysis patients who have not received any FIR therapy within the previous 12 months
* Patients on a standard continuous ambulatory peritoneal dialysis (CAPD) (1.5-2 L; 4-5 exchanges/day) or ambulatory peritoneal dialysis (APD) program

Exclusion Criteria:

* History of CAPD-related peritonitis within 3 months prior to the study period;
* History of cerebrovascular accident or myocardial infarction or interventional procedure (percutaneous transluminal coronary angioplasty or stent) for coronary artery disease within the 3 months prior to the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
KT/V | Change from baseline level at 6 months and 12 months
  K - dialyzer urea clearance; t - dialysis time; V - total volume within the body that urea is distributed
Weekly creatinine clearance | Change from baseline level at 6 months and 12 months
  WCCr (L/wk/1.73m^2)

SECONDARY OUTCOMES:
Ultrafiltration volume | Change from baseline level at 6 months and 12 months
  Peritoneal function parameter (mL)
Net volume | Change from baseline level at 6 months and 12 months
  Peritoneal function parameter (mL)
D/D0 glucose ratio | Change from baseline level at 6 months and 12 months
  Peritoneal function parameter
D/PCr ratio | Change from baseline level at 6 months and 12 months
  Peritoneal function parameter
D/P urea ratio | Change from baseline level at 6 months and 12 months
  Peritoneal function parameter
Albumin | Change from baseline level at 6 months and 12 months
  Biochemical function parameter (g/dL)
Blood urea nitrogen | Change from baseline level at 6 months and 12 months
  Biochemical function parameter (mg/dL)
Creatinine | Change from baseline level at 6 months and 12 months
  Biochemical function parameter (mg/dL)
Major cardiovascular adverse events | Change from baseline level at 12 months
  3-point major adverse cardiovascular events (3P-MACE) comprising of non-fatal stroke, myocardial infarction, and cardiovascular death, coronary artery disease (CAD), hospitalized heart failure (HHF)
Infection events (number of hospital admission events) | Change from baseline level at 12 months
  Pneumonia, peritonitis

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Ching Lin, MD, PhD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lin CC, Chang CF, Lai MY, Chen TW, Lee PC, Yang WC. Far-infrared therapy: a novel treatment to improve access blood flow and unassisted patency of arteriovenous fistula in hemodialysis patients. J Am Soc Nephrol. 2007 Mar;18(3):985-92. doi: 10.1681/ASN.2006050534. Epub 2007 Jan 31. PMID 17267744
- [Background] Lin CC, Liu XM, Peyton K, Wang H, Yang WC, Lin SJ, Durante W. Far infrared therapy inhibits vascular endothelial inflammation via the induction of heme oxygenase-1. Arterioscler Thromb Vasc Biol. 2008 Apr;28(4):739-45. doi: 10.1161/ATVBAHA.107.160085. Epub 2008 Jan 17. PMID 18202320
- [Background] Lin CC, Yang WC, Chen MC, Liu WS, Yang CY, Lee PC. Effect of far infrared therapy on arteriovenous fistula maturation: an open-label randomized controlled trial. Am J Kidney Dis. 2013 Aug;62(2):304-11. doi: 10.1053/j.ajkd.2013.01.015. Epub 2013 Mar 6. PMID 23474008
- [Background] Lin CC, Chung MY, Yang WC, Lin SJ, Lee PC. Length polymorphisms of heme oxygenase-1 determine the effect of far-infrared therapy on the function of arteriovenous fistula in hemodialysis patients: a novel physicogenomic study. Nephrol Dial Transplant. 2013 May;28(5):1284-93. doi: 10.1093/ndt/gfs608. Epub 2013 Jan 22. PMID 23345623